CLINICAL TRIAL: NCT03808727
Title: Massed Cognitive Processing Therapy for Combat-related PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Boston Healthcare System (U.S. Federal Agency)
Collaborators: Fort Belvoir Community Hospital (U.S. Federal Agency); The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Jennifer Schuster Wachen, Ph.D., Principal Investigator, VA Boston Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: W81XWH-17-2-0067
Record Dates: First submitted 2019-01-16; First posted 2019-01-18 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: PTSD, Post Traumatic Stress Disorder
Keywords: cognitive processing therapy; CPT; PTSD; military
MeSH Terms: conditions — Combat Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Massed Cognitive Processing Therapy (MCPT) (Experimental): Cognitive Processing Therapy is an evidence-based form of Cognitive Behavioral Therapy (CBT) used to treat PTSD. CPT is a 12-session manualized program that focuses on challenging beliefs and assumptions related to the trauma, oneself, and the world. MCPT will be delivered in an intensive outpatient setting (12 sessions in 5 days) composed of both group and individual sessions.
  Interventions: Behavioral: Cognitive Processing Therapy
- Standard Cognitive Processing Therapy (Active Comparator): Cognitive Processing Therapy is an evidence-based form of Cognitive Behavioral Therapy (CBT) used to treat PTSD. CPT is a 12-session manualized program that focuses on challenging beliefs and assumptions related to the trauma, oneself, and the world. Standard CPT will be delivered in 12 one-hour sessions over 6 weeks and involves only individual sessions.
  Interventions: Behavioral: Cognitive Processing Therapy

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy — Cognitive Processing Therapy is an evidence-based form of Cognitive Behavioral Therapy (CBT) used to treat PTSD. CPT is a 12-session manualized program that focuses on challenging beliefs and assumptions related to the trauma, oneself, and the world.

SUMMARY:
The purpose of this study is to determine if cognitive processing therapy (CPT) delivered in a massed format (MCPT) is as effective as standard delivery of CPT. MCPT will be delivered in an intensive outpatient setting (12 sessions in 5 days) composed of both group and individual sessions. Standard delivery of CPT consists of 12 sessions over 6 weeks and involves only individual sessions. Assessment of PTSD and related symptoms will be conducted at pre-treatment and 1 month and 4 months following treatment in both conditions. Additionally, in order to compare the treatment groups at the same point in actual time, each group will be assessed at the one month posttreatment time point for the other condition.

DETAILED DESCRIPTION:
Cognitive Processing Therapy (CPT) is identified as one of the most effective treatments for posttraumatic stress disorder (PTSD) in a wide range of trauma populations, with a higher effect size than any other evidence-based treatments for PTSD. However, CPT has been shown to be somewhat less effective in active duty and veteran populations when compared to civilian trauma victims. One reason may be that service members have difficulty committing to a six-week course of therapy due to the demanding nature of active duty military operations schedules. In addition, limited availability of clinical providers may reduce access to care. One way to address these barriers may be to administer CPT in an intensive, 5-day format. This format may increase rates of treatment completion and produce faster symptom improvement than the standard administration of CPT. This study will test the efficacy of massed CPT (MCPT) compared to standard CPT delivery. MCPT will be delivered in an intensive outpatient setting (12 sessions in 5 days) composed of both group and individual sessions. Standard delivery of CPT consists of 12 sessions over 6 weeks and involves only individual sessions.

The sample includes 140 active duty service members randomized to receive either MCPT or standard CPT. Participants will be assessed 4 times during the course of the study. In order to test the equivalence of the treatment conditions, outcomes will be compared at a consistent number of weeks posttreatment for each condition (e.g., at baseline, and one month and 4 months following the conclusion of the therapy). Additionally, in order to compare the treatment groups at the same point in actual time, each group will be assessed at the one month posttreatment time point for the other condition. The timing of these assessment intervals allows for the comparison groups to be assessed similarly at each important juncture of therapy (baseline and post-treatment) and also to be assessed for maintenance of treatment gains following a similar passage of time (4 months post-treatment). Those who drop out of treatment will be asked to return for the follow-up assessments based on their projected end date for inclusion in the intent to treat analyses.

Aim 1: To evaluate the efficacy of massed CPT in a sample of active duty military in reductions of clinician-rated and self-reported PTSD symptoms, as well as secondary outcomes including depression, psychosocial functioning, and physical health after treatment completion (assessed at one month and 4 months posttreatment for each condition). Rates of treatment completion and speed of recovery will also be compared between conditions.

Aim 2: To examine predictors of symptom reduction in each treatment condition including demographic characteristics, military factors, psychosocial variables, and comorbid mental health symptoms.

Aim 3 (Exploratory): To evaluate the tolerability of massed versus standard administration of CPT. Important nonspecific factors such as therapeutic alliance, patient preference, treatment expectancy, perceived burden, and emotional factors such as anxiety and avoidance will be examined with regard to treatment outcome.

To test the hypotheses regarding noninferiority of the MCPT treatment condition relative to CPT, 95% conﬁdence interval (CI) on the difference in CAPS scores (and other measures) between conditions will be constructed for each measurement period. MCPT will be deemed noninferior to CPT, thus supporting hypotheses 1 and 2 if the upper limit of the CI is less than 10 for CAPS - the a priori specified noninferiority margin.

To examine differences in treatment completion between conditions, frequencies (and proportions) in a chi-square test of independence will be used. That is, if 70 participants begin the study in each condition, the proportion that drops out prior to completion of treatment is expected to be significantly less in the MCPT condition. To examine speed of recovery, scores on outcomes at 5 weeks from baseline (one month post treatment for MCPT, mid-treatment for CPT) will be compared via an a priori specified t-test.

In addition, a multilevel approach to analyzing longitudinal data 95 using the Linear and Nonlinear Mixed Effects Models package from 96 will be utilized for further tests and exploration of changes in measures of PTSD and secondary outcomes. Multilevel modeling is ideal for studies which employ repeated measurements nested within individuals such as is the case in this design. To examine individual predictors of symptom reduction (Aim 2), the four measurement occasions will be leveraged to assess both group and individual differences in trajectories for each of the study outcomes. Individual difference variables will be added to the models as moderators of condition and time (i.e., to what extent do change patterns vary by these individual variables?). For Aim 3, a similar strategy will be used but leveraging the nonspecific factors as the outcomes and session as the time variable. Thus, the extent to which nonspecific factors change as a function of treatment condition over the sessions will be examined.

Lastly, an additional one-year follow-up assessment was added as an exploratory aim to examine longer-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female (age 18+) active duty military seeking treatment for PTSD
* Diagnosis of PTSD determined by a clinician-administered Posttraumatic Stress Scale (CAPS-5)
* Speak and read English

Exclusion Criteria:

* Current suicide or homicide risk meriting crisis intervention
* Active psychosis
* Moderate to severe brain damage (as determined by the inability to comprehend the baseline screening questionnaires)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in PTSD symptoms as assessed by the Clinician Administered PTSD Scale (CAPS-5) | Baseline, one-month posttreatment, 4 months posttreatment (weeks 0, 5, 10, 17, 22, depending on tx condition)
  The CAPS is a semi-structured interview to assess presence and severity of PTSD symptoms. The total score on the CAPS will be used as the primary outcome measure in this study.
Change in PTSD symptoms as assessed by the PTSD Check List - DSM-5 (PCL-5) | Baseline, one-month posttreatment, 4 months posttreatment (weeks 0, 5, 10, 17, 22, depending on tx condition) and weekly or daily during treatment
  The PCL-5 is a 20-item self-report measure based upon the Diagnostic and Statistical Manual (DSM-5) criteria for PTSD

SECONDARY OUTCOMES:
Change in depressive symptoms as measured by the Patient Health Questionnaire-9 (PHQ-9) | Baseline, one-month posttreatment, 4 months posttreatment (weeks 0, 5, 10, 17, 22, depending on tx condition) and weekly or daily during treatment
  The PHQ-9 is a widely used and well-validated instrument for measuring the severity of depressive symptoms
Change in suicidality as measured by the Depressive Symptom Index - Suicidality Subscale (DSI-SS) | Baseline, one-month posttreatment, 4 months posttreatment (weeks 0, 5, 10, 17, 22, depending on tx condition) and weekly or daily during treatment
  The DSI-SS is a 4-item self-report measure of suicidal ideation that focuses on ideation, plans, perceived control over ideation, and impulses for suicide.
Changes in functioning as measured by the Well-Being Inventory (WBI) | Baseline, one-month posttreatment, 4 months posttreatment (weeks 0, 5, 10, 17, 22, depending on tx condition)
  The WBI provides a multidimensional assessment of status, functioning, and satisfaction in the four key life domains of vocation, finances, health, and social relationships.This study will only include the subscales measuring functioning and satisfaction in the domains of work, health, and social relationships.
Changes in alcohol use as measured by the Alcohol Use Disorders Identification Test (AUDIT) | Baseline, one-month posttreatment, 4 months posttreatment (weeks 0, 5, 10, 17, 22, depending on tx condition)
  The AUDIT is a 10-item screening measure, developed by the World Health Organization (WHO), with three subscales (alcohol consumption, drinking behavior, and alcohol-related problems)
Changes in anger as measured by the Dimensions of Anger Reactions-5 (DAR-5) | Baseline, one-month posttreatment, 4 months posttreatment (weeks 0, 5, 10, 17, 22, depending on tx condition)
  The DAR-5 63 is a short form version of the original Dimensions of Anger Reactions. 64 It addresses anger frequency, intensity, duration, aggression, and interference with social functioning.
Changes in health functioning as measured by the Veterans Rand 12-Item Health Survey (VR-12) | Baseline, one-month posttreatment, 4 months posttreatment (weeks 0, 5, 10, 17, 22, depending on tx condition)
  The Veterans VR-12 was developed from the Veterans VR-36 and adapted from the Short Form -36 (SF-36), and spans the range of health domains from physical to psychological health status.
Change in somatic symptoms as measured by the Patient Health Questionnaire - 15 (PHQ-15) | Baseline, one-month posttreatment, 4 months posttreatment (weeks 0, 5, 10, 17, 22, depending on tx condition)
  The PHQ-15 70 is an abbreviated version of the original PHQ that asks about somatic symptoms and symptom clusters
Change in sleep disturbance as measured by the Insomnia Severity Index (ISI) | Baseline, one-month posttreatment, 4 months posttreatment (weeks 0, 5, 10, 17, 22, depending on tx condition)
  The ISI is a 7-item self-report measure that assesses perceived severity of insomnia.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Wachen, Ph.D., Principal Investigator — VA Boston Healthcare System
Locations (1):
- Fort Belvoir Community Hospital, Fort Belvoir, Virginia, United States